CLINICAL TRIAL: NCT02574039
Title: Absorption, Metabolism and Excretion of Oat Phenolic Acids in Healthy Men.
Brief Title: Oat Phenolics Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PROGRAIN1
Record Dates: First submitted 2015-06-26; First posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: volunteers; oat; phenolic acid; bioavailability
MeSH Terms: conditions — Gyrate Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oat bran (Experimental): 66g oat bran made up in 350ml skimmed milk
  Interventions: Dietary Supplement: Oat bran
- Control (Placebo Comparator): Refined grain product and 350ml skimmed milk
  Interventions: Dietary Supplement: refined grain

INTERVENTIONS:
Dietary Supplement: Oat bran — 66g oat bran made up in 350ml skimmed milk
  Arms: Oat bran
Dietary Supplement: refined grain — refined grain product and 350ml skimmed milk
  Arms: Control

SUMMARY:
A diet rich in whole grain is inversely associated with cardiovascular disease risk and this benefit could be partly attributed to the phenolic acid content of whole grains. The exact absorption, metabolism and excretion of whole grain phenolic acids, however, is not fully understood. In a small human intervention trial, the investigators will investigate to what extent phenolic acids from whole grain oats are absorbed, excreted in urine and how they are metabolised.

ELIGIBILITY:
Inclusion Criteria:

* Males
* 25 to 65 years old

Exclusion Criteria:

* Allergies to oats
* Parallel participation in another research project
* Having flu vaccination or antibiotics within 3 months of trial start
* Taking food supplements within 3 months of trial start
* Past or existing medical history of vascular disease, diabetes, hepatic, renal, gastrointestinal, haematological, neurological, thyroidal disease or cancer

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in phenolic acid metabolite excretion | Baseline and 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food and Nutritional Sciences, Reading, Berkshire, United Kingdom